CLINICAL TRIAL: NCT01423097
Title: Magnitude of Osteoarthritis disadVantage on pEoples liveS
Acronym: MOVES
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RPO-XXX-2011/2
Record Dates: First submitted 2011-08-24; First posted 2011-08-25 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis symptoms
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Estimate the prevalence of self-reported osteoarthritis and its characterization in adults over 45 years of age:

* Characterization of self-reported patients with OA (socio-demographic, comorbidities, VAS for intensity of pain)
* Characterization of OA diagnosis in patients with self-reported OA
* Impact of self-reported OA in the working abilities, quality of life and functionality (SF-12 v2.0)
* Characterization of treatment approaches (therapeutic and non-therapeutic) for self-reported patients with OA
* Patient perception of impact of OA in its life and importance given to disease

DETAILED DESCRIPTION:
Magnitude of Osteoarthritis disadvantage on peoples lives.

ELIGIBILITY:
Inclusion Criteria:

- Adults over 45 years old with self-reported osteoarthritis

Exclusion Criteria:

- NA

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Estimate the prevalence of self-reported osteoarthritis (OA) in adults over 45 years of age by direct interview. | Single interview at the only one patient contact

SECONDARY OUTCOMES:
Characterization of self-reported patients with OA by collecting socio-demographic information through direct interview. | Single interview at the only one patient contact
Characterization of self-reported patients with OA by collecting comorbidities information through direct interview. | Single interview at the only one patient contact
Characterization of self-reported patients with OA by collecting information for intensity of pain through direct interview. | Single interview at the only one patient contact
Characterization of OA diagnosis in patients with self-reported OA by direct interview. | Single interview at the only one patient contact
Impact of self-reported OA in the working abilities, quality of life and functionality using Questionnaire SF-12 v2.0 | Single interview at the only one patient contact
Patient perception of impact of OA in its life and importance given to disease by direct interview. | Single interview at the only one patient contact

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Queluz Baixo, Barcarena, Portugal